CLINICAL TRIAL: NCT03771560
Title: An Examination of Changes in Urinary Metabolites With Use of Folinic Acid in Children With Autism Spectrum Disorder (ASD)
Brief Title: Folinic Acid in Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Robert Hendren, Professor of Psychiatry, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Folinic acid
Record Dates: First submitted 2018-02-14; First posted 2018-12-11 (Actual); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): In this open-label trial, all subjects will receive the twice daily dose of folinic acid. Folinic acid will be delivered in pill form at a weight-based dose.
  Interventions: Drug: folinic acid

INTERVENTIONS:
Drug: folinic acid — subject will take folinic acid daily for 12 weeks
  Other Names: leucovorin calcium

SUMMARY:
An examination of changes in urinary metabolites with use of folinic acid in children with autism spectrum disorder (ASD). Investigators will also measure behavioral measures and academic measures monthly at school with teachers and parents report.

DETAILED DESCRIPTION:
Children enrolled in Oak Hill School will enroll in this study and take folinic acid supplement twice a day for 12 weeks period. Behavioral measures and urinary metabolites will be collected pre and post treatment. Behavioral measures will be taken again at 16 weeks, after 4 weeks of not dosing.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 5 and 25

Exclusion Criteria:

* Not currently taking folinic acid

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Folinic Acid Open-label: In this open-label trial, all subjects will receive the twice daily dose of folinic acid. Folinic acid will be delivered in pill form at a weight-based dose.
  folinic acid: subject will take folinic acid daily for 12 weeks
Period: Overall Study
Arm/Group | Folinic Acid Open-label
Started | 18
Completed | 12
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Children with ASD enrolled in Oak Hill school and completed the entire study.
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 16 [13 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 3
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist (ABC) - Parent Reported Change
Description: The Aberrant Behavior Checklist - parent reported version measures aberrant behavior in children and young adults. There are 58 questions.The scoring of one question can range from 0 (not a problem) to 3 (severe) points on a Likert scale. The total possible score range for the ABC is 0 - 174. Analysis will be performed for mean of total score change over time.
  Scoring from 0-3
  Not a problem = 0, Slightly = 1, Moderately Serious =2, Severe =3
  Lower score indicates better performance.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 12
score on a scale | -2.4 [-11.3 to 6.4]
Statistical Analysis 1: Comparison: Folinic Acid Open-label; The parent-reported change in mean ABC total score from baseline to week 12; Test type: Other; p = 0.56, Paired Sample t-test; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-11.3 to 6.4]

2. Primary Outcome: Aberrant Behavior Checklist (ABC) - Teacher Reported Change
Description: The Aberrant Behavior Checklist - teacher reported version measures aberrant behavior in children and young adults. There are 58 questions. The scoring of ABC questions can range from 0 (not a problem) to 3 (severe) points on a likert scale. The total possible score range for the ABC is 0 - 174. Analysis will be performed for mean of total score change over time.
  Scoring from 0-3
  Not a problem = 0, Slightly = 1, Moderately Serious =2, Severe =3
  Lower score indicates better performance.
Time Frame: Baseline to Week 12
Population: Deleted one outlier for data analysis; deleted one subject because of missing survey time point from teacher.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 10
score on a scale | 1.2 [-5.2 to 7.6]
Statistical Analysis 1: Comparison: Folinic Acid Open-label; The teacher-reported change in mean ABC total score from baseline to week 12; Test type: Other; p = 0.68, Paired Sample t-test; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-5.2 to 7.6]

3. Secondary Outcome: Social Responsiveness Scale (SRS) - Parent Reported Change
Description: The Social Responsiveness Scale - parent reported version measures social ability in children and young adults. There are 65 questions. The questions on the scale with anchors 1 (Not True) - 4 (Almost Always True). The scoring of SRS questions can range from 0-3 (with possible reverse scoring) based on scoring instructions for data analysis. The total possible score range for the SRS is 0 - 195. Analysis will be performed for mean of total score change over time.
  Anchors Not True = 1 Sometimes True = 2 Often True = 3 Almost Always True = 4
  Lower score indicates better performance.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 12
score on a scale | -7.8 [-17.3 to 1.6]
Statistical Analysis 1: Comparison: Folinic Acid Open-label; The parent-reported change in mean SRS total score from baseline to week 12; Test type: Other; p = 0.095, Paired Sample t-test; Mean Difference (Final Values) = -7.8, 95% CI 2-sided [-17.3 to 1.6]

4. Secondary Outcome: Social Responsiveness Scale (SRS) - Teacher Reported Change
Description: The Social Responsiveness Scale - teacher reported version measures social ability in children and young adults. There are 65 questions. The questions on the scale with anchors 1 (Not True) - 4 (Almost Always True). The scoring of SRS questions can range from 0-3 (with possible reverse scoring) based on scoring instructions for data analysis. The total possible score range for the SRS is 0 - 195. Analysis will be performed for mean of total score change over time.
  Anchors Not True = 1 Sometimes True = 2 Often True = 3 Almost Always True = 4
  Lower score indicates better performance.
Time Frame: Baseline to Week 12
Population: Deleted one outlier for data analysis; deleted one subject because of missing survey time point from teacher.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 10
score on a scale | -0.5 [-7.0 to 13.5]
Statistical Analysis 1: Comparison: Folinic Acid Open-label; The teacher-reported change in mean SRS total score from baseline to week 12; Test type: Other; p = 0.95, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.5, 95% CI 2-sided [-7.0 to 13.5]

5. Secondary Outcome: Pediatric Quality of Life (PedsQL) - Parent Reported Change
Description: Pediatric Quality of Life is reported by parent only and it assesses improvement of the child's overall quality of life through questions about physical, emotional, social and school functioning. There are 23 questions. The scoring of PedsQL questions can range from 0 (Never) to 4 (Almost Always) points on a Likert scale. Questions are reversed scored and linearly transformed to a 0 - 100 scale for data analysis as follows: 0=100, 1=75, 2=50, 3=23, 4=0. The total score = sum of all the questions over the number of items answered on. The total possible score range for the PedsQL is 0 - 100. Analysis will be performed for mean of total score change over time.
  Scoring from 0 to 4
  Never = 0, Almost Never = 1, Sometimes = 2, Often = 3, Almost Always =4
  Higher score indicates better performance.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Folinic Acid Open-label
Number analyzed (Participants) | 12
score on a scale | -0.8 [-5.2 to 3.5]
Statistical Analysis 1: Comparison: Folinic Acid Open-label; The parent-reported change in mean PedsQL total score from baseline to week 12; Test type: Other; p = 0.69, Paired Sample t-test; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.2 to 3.5]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Folinic Acid Open-label
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folinic Acid Open-label (N=12)
Upset Stomach (Gastrointestinal disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased aggression (Psychiatric disorders) | 1 (1)
Blood in Stool (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT03771560/Prot_SAP_000.pdf